CLINICAL TRIAL: NCT02293499
Title: Peer Led Asthma Self Management for Adolescents: PLASMA
Acronym: PLASMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Johns Hopkins University (Other); University of Tennessee (Other)
Responsible Party: Principal Investigator, Hyekyun Rhee, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSRB00053987
Record Dates: First submitted 2014-10-24; First posted 2014-11-18 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Asthma
Keywords: asthma; adolescent; intervention
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Masking Description: Given the overt nature of the intervention, blinding either participants or investigators was not achieved although we did not inform participants of their group membership explicitly.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peer Led Asthma Self-Management (Active Comparator): Peer-led asthma self-management for adolescents : PLASMA will be implemented in small groups at a camp setting where paired peer-leaders will facilitate learning activities.Paired peer leaders will share and coordinate the responsibilities of facilitating group activities. Training content includes: Day 1: Asthma basics and prevention; Day 2: Asthma monitoring and management; Day 3: Communication/ psychosocial issue management/leadership training/hands-on practice in simulated peer-led group settings (role-play)
  Interventions: Behavioral: PLASMA
- Adult Led Asthma Self-Management (Active Comparator): The adult led asthma self-management will take place within 2 weeks of the peer-led camp to minimize the history effect. Two healthcare professionals will attend peer-leader training sessions to become familiar with the program content, then lead instructional activities. As in PLASMA, adult leaders will base their instruction on the program manual to ensure comparable program content. Adult leaders will adopt mainly a didactic format and skill demonstration.
  Interventions: Behavioral: PLASMA

INTERVENTIONS:
Behavioral: PLASMA — A structured asthma self-management manual ("Let's Talk about Asthma [LTAA],"developed by the study team will be utilized in a camp like setting and administered by either peers or adults medical professionals. The manual adheres to the 2007 NAEPP Guidelines Training strategies will involve didactic sessions, discussion, demonstrations, and role-play. Group learning activities will closely align with the program manual (LTAA) that consists of three sessions. Participants will also learn and practice skills in using the peak flow meter, spacer and inhaler, daily symptom diary and asthma action plan. Besides instructional activities, participants will engage in recreational activities that each camp site.

SUMMARY:
Asthma is a serious chronic health condition particularly in inner-city adolescents, who suffer disproportionately high asthma-related morbidity and mortality that place heavy economic burdens on families and society. There is a consensus that adverse asthma outcomes can be ameliorated by an individual's active engagement in adequate self-management. This multi-site randomized controlled study proposes to implement and evaluate a peer-led asthma self-management for adolescents (PLASMA) program that has demonstrated its feasibility and preliminary efficacy in a previous study. PLASMA will be implemented in three cities (Buffalo NY, Baltimore MD, and Memphis TN) that have particularly high rates of pediatric asthma and asthma-related morbidity, and are thus most likely to benefit from the program. PLASMA comprises three main components: (a) peer-leader training; (b) a one-day asthma camp where peer leaders will deliver manualized self-management content recommended by the national guidelines; and (c) bi-monthly peer-leader contacts. Specific aims are: (1) to evaluate the effectiveness of PLASMA in inner-city adolescents with asthma in improving quality of life (primary outcome), and asthma knowledge, attitudes, outcome expectations, self-efficacy, self-management skills, and asthma control, FEV1 (exploratory outcomes) over time, compared to a control group for whom adult leaders will deliver the same program content; (2) to examine the mediating effects of the exploratory outcomes on quality of life; (3) to examine the moderating effects of personal factors (e.g., age, sex, family support) on the intervention's primary and exploratory outcomes; (4) to evaluate the effects of PLASMA on study outcomes in peer leaders (16-20 years); and (5) to determine the economic impact of the intervention. These aims will be accomplished using a two-group randomized controlled trial with 378 adolescents (12-17 years) from the three cities (126 for each site). A total of 42 qualified peer leaders (14 in each site) will be enrolled based on adult nomination. Eligibility criteria for both peer leaders and adolescent learners include: a current asthma diagnosis; persistent asthma; absence of other chronic or mental illness; inner-city residence; and capability of verbal and written communication in English. Participants will provide data at enrollment (T1), camp (T2), and at 3-, 6-, 9-, 12-, and 15-months post-camp (T3-T7). Data will be analyzed using a multi-site hierarchical three-level linear mixed-effects model where level 1 represents repeated measures, level 2 = subject, and level 3 = site. To determine the economic impact of the program, investigator will measure the direct healthcare costs and total costs of the program, and perform net cost analyses for each type of costs. In addition, investigator will estimate cost-effectiveness ratios of the PLASMA group compared with the control.

DETAILED DESCRIPTION:
Asthma, the most common pediatric chronic condition, is a serious problem for many adolescents. In 2010, nearly 11% of adolescents (2.7 million) ages 12 through 17 years in the US reported current asthma. This age cohort suffers greater asthma-related morbidity and mortality than younger children. Asthma disproportionately affects inner-city youth, where asthma severity has increased and achieving optimum asthma control has been elusive. Several factors including poor socioeconomic conditions, life stresses, and environmental triggers have been found to be associated with poorly controlled asthma in inner-city children. Programs targeting asthma in inner-city children have primarily focused on the modification of environmental factors and addressing disparity in healthcare access. Limited intervention efforts have been directed to address high inner-city asthma morbidity specifically in adolescents by promoting adequate self-management.

Dr. Rhee successfully completed an R21 (NR009837) where she designed an evidence-based peer-led asthma self-management for adolescents (PLASMA) program and tested its efficacy in a randomized parallel group design in 112 urban and suburban adolescents with persistent asthma. The PLASMA program was implemented at a one-day camp and involved monthly follow-ups by peer leaders. The program was well received by participants, and relative to adolescents who received an adult-led program, the PLASMA group reported better quality of life and asthma control and fewer asthma-related urgent office visits. Subgroup analysis revealed that the program was particularly effective for inner-city adolescents in improving asthma outcomes compared with suburban participants. Given the disproportionate burdens of asthma in inner-city youth and the program's compelling effects in this population, focusing on inner-city adolescents as a target of the PLASMA program is critical.

Building on this previous trial of efficacy, the overall goal of the proposed study is to evaluate the effectiveness and generalizability of the peer-led intervention, PLASMA, in improving asthma outcomes in inner-city adolescents from three metropolitan cities in the Northern, Eastern and Southern US with distinctive historical and cultural backgrounds. Multisite studies have been advocated as an effective approach to strengthening external validity as such studies afford the opportunity to assess the extent to which treatment effects are generalizable to different settings. Ascertaining generalizability across sites is important as it guides future translation of study findings into policy and practice. This study will also determine long-term sustainability of PLASMA effects and estimate the economic impact of the intervention. This multi-site study is significant in that it will target the understudied population, inner-city adolescents with asthma in three cities in the US, who present serious challenges to optimum asthma management.

Specific study aims are:

1. To evaluate systematically the effectiveness of a peer-led asthma program in inner-city adolescents with persistent asthma. This aim will be accomplished by using a two-group randomized controlled trial with 378 adolescents (12-17 years) from the three cities. The intervention group will receive PLASMA involving peer leader training, a one-day intense asthma self-management program led by peer leaders and bimonthly contacts from peer leaders. Intervention effects will be examined in comparison to the control group, who will receive the same program content delivered by adult leaders. Investigators hypothesize that: relative to the control group, the PLASMA group will report greater improvement over time in (H1) quality of life (primary outcome), and (H2) asthma knowledge, attitudes, outcome expectations, self-efficacy, self-management skills, and asthma control, FEV1 (exploratory outcomes). (H3) The post-PLASMA scores on outcome measures will be higher than pre-program scores from both treatment groups.
2. To examine the mediating effects of the secondary outcomes (knowledge, attitudes, outcome expectations, self-efficacy, self-management skills, asthma control, and FEV1) on the primary outcome (quality of life) of the intervention.
3. To examine the moderating effects of personal factors (e.g., age, sex, family support) on primary and secondary outcomes of the intervention.
4. To evaluate the effects of PLASMA on primary and exploratory outcomes in peer leaders (16-20 years). Investigators hypothesize that the peer leaders (n=42) will report significant improvement in quality of life (primary outcome) and secondary outcomes (knowledge, attitudes, outcome expectations, self-efficacy, self-management skills, asthma control and FEV1) over the course of 15 months.
5. To determine the economic impact of the intervention. This aim will be accomplished by (5a) measuring the direct healthcare costs and total costs of the PLASMA program, as compared with the control group; (5b) performing net cost analyses for each type of costs; and (5c) estimating cost-effectiveness ratios of the PLASMA group compared with the control. Investigators hypothesize that the direct and overall costs per participant in the PLASMA group will be less than costs per participant in the control group, or cost neutral.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria for adolescent (camp) participants include:

  1. age between 12-17 years;
  2. physician-diagnosed asthma that has required health service use (preventive or acute) within 12 months prior to recruitment;
  3. persistent asthma determined by current use of a control medication or presenting at least one of the following four symptom levels in the past 4 weeks, as defined by the NAEPP guidelines91:
* > 2 days/week of daytime symptoms,
* >3-4 times of nighttime awakening,
* >2 days/week of SABA use, or
* any interference with normal activities due to asthma (4) Investigators will include those with chronic health conditions except for those with conditions affecting respiratory system, heart disease, pneumonia, etc., and those with moderate to severe cognitive impairments; (5) primary residence located in the participating inner cities based on zip codes; and (6) ability to understand spoken and written English.

Eligibility criteria for peer leaders include:

1. age between 16-20 years;
2. nomination from school teachers/nurses or healthcare providers for candidates' exemplary asthma self-management, leadership, and emotional intelligence; and
3. fulfillment of eligibility criteria (2)-(6) prescribed for adolescent participants.

Exclusion Criteria:

1. Adolescents who are pregnant or incarcerated at enrollment;
2. Have learning disabilities based on reports from teachers or clinicians will be excluded from the study because such conditions can confound the interpretation of findings;
3. Those who have serious health (other than asthma) and emotional preconditions (e.g., severe depression, anxiety disorders, schizophrenia).

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 371 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - University at Buffalo, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of Tennessee, Memphis, Tennessee

REFERENCES:
- [Derived] Rhee H, Love T, Wicks MN, Tumiel-Berhalter L, Sloand E, Harrington D, Walters L. Long-term Effectiveness of a Peer-Led Asthma Self-management Program on Asthma Outcomes in Adolescents Living in Urban Areas: A Randomized Clinical Trial. JAMA Netw Open. 2021 Dec 1;4(12):e2137492. doi: 10.1001/jamanetworkopen.2021.37492. PMID 34874404
- [Derived] Rhee H, Love T, Mammen J. Comparing Asthma Control Questionnaire (ACQ) and National Asthma Education and Prevention Program (NAEPP) asthma control criteria. Ann Allergy Asthma Immunol. 2019 Jan;122(1):58-64. doi: 10.1016/j.anai.2018.09.448. Epub 2018 Sep 11. PMID 30213611
- [Derived] Rhee H, Love TM, Harrington D, Grape A. Comorbidity of atopy in urban adolescents with asthma. Ann Allergy Asthma Immunol. 2017 Nov;119(5):466-467. doi: 10.1016/j.anai.2017.08.017. No abstract available. PMID 29150074

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 446 screened participants, 320 met eligibility criteria and were enrolled and randomized to one of the two arms. Of 72 screened peer-leaders, 51 met criteria and were enrolled as peer-leaders as outlined in the intervention arm of the study, for a total of 371 enrolled individuals.
Groups:
- Adult Led Asthma Self-Management: PLASMA: A structured asthma self-management manual ("Let's Talk about Asthma [LTAA],"developed by the study team will be utilized in a camp like setting and administered by either peers or adults medical professionals. The manual adheres to the 2007 NAEPP Guidelines Training strategies will involve didactic sessions, discussion, demonstrations, and role-play. This arm is the adult-led control group.
- Peer Led Asthma Self-Management: PLASMA: A structured asthma self-management manual ("Let's Talk about Asthma [LTAA],"developed by the study team will be utilized in a camp like setting and administered by either peers or adults medical professionals. The manual adheres to the 2007 NAEPP Guidelines Training strategies will involve didactic sessions, discussion, demonstrations, and role-play. This arm is the peer-led intervention group.
- Peer Leaders: PLASMA: A structured asthma self-management manual ("Let's Talk about Asthma [LTAA],"developed by the study team will be utilized in a camp like setting and administered by either peers or adults medical professionals. The manual adheres to the 2007 NAEPP Guidelines Training strategies will involve didactic sessions, discussion, demonstrations, and role-play. This group is the peer leaders who facilitated the Peer--led intervention group intervention.
Period: Baseline - Enrollment
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Started | 152 | 168 | 51
Completed | 152 | 168 | 51
Not Completed | 0 | 0 | 0
Period: Training - Peer Leaders Only
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Started (Only the Peer leader arm of this study participated in this time point by study design.) | 0 (Participant number carried over from previous time point.) | 0 (Participant number carried over from previous time point.) | 51
Completed | 0 | 0 | 41
Not Completed | 0 | 0 | 10
Not completed — By design, two treatment groups did not participate; 10 peer leaders were Withdrawn by PI | 0 | 0 | 10
Period: Intervention - Camp
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Started | 152 (By design, they did not participate in the previous period.) | 168 (By design, they did not participate in the previous period.) | 41
Completed | 125 | 134 | 35
Not Completed | 27 | 34 | 6
Not completed — Withdrawal by Subject | 3 | 6 | 2
Not completed — these are those not showing up at camp | 24 | 28 | 4
Period: 3 Month Follow Up
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Started | 149 | 162 | 39
Completed | 134 | 147 | 29
Not Completed | 15 | 15 | 10
Not completed — Withdrawal by Subject | 1 | 0 | 4
Not completed — Lost to Follow-up | 14 | 15 | 6
Period: 6 Month Follow Up
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Started | 148 | 162 | 35
Completed | 131 | 135 | 28
Not Completed | 17 | 27 | 7
Not completed — Lost to Follow-up | 17 | 27 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: 9 Month Follow Up
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Started | 148 | 162 | 34
Completed | 122 | 134 | 30
Not Completed | 26 | 28 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Lost to Follow-up | 24 | 28 | 4
Period: 12 Month Follow Up
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Started | 146 | 162 | 34
Completed | 120 | 136 | 28
Not Completed | 26 | 26 | 6
Not completed — Lost to Follow-up | 26 | 25 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: 15 Month Follow Up
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Started | 146 | 161 | 34
Completed | 124 | 139 | 27
Not Completed | 22 | 22 | 7
Not completed — Lost to Follow-up | 22 | 22 | 7

BASELINE CHARACTERISTICS:
Groups:
- Peer Led Asthma Self-Management: PLASMA: A structured asthma self-management manual ("Let's Talk about Asthma [LTAA],"developed by the study team will be utilized in a camp like setting and administered by either peers or adults medical professionals. The manual adheres to the 2007 NAEPP Guidelines Training strategies will involve didactic sessions, discussion, demonstrations, and role-play. This arm is the peer--led intervention group.
- Total: Total of all reporting groups
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders | Total
Number analyzed (Participants) | 152 | 168 | 51 | 371
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.19 (1.647) | 14.33 (1.750) | 17.22 (1.270) | 14.67 (1.935)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 78 | 33 | 185
  Male | 78 | 90 | 18 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 13 | 1 | 31
  Not Hispanic or Latino | 135 | 155 | 50 | 340
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 21 | 23 | 11 | 55
  African American/Black | 120 | 131 | 40 | 291
  American Indian/Alaska Native | 2 | 1 | 0 | 3
  Asian | 0 | 1 | 0 | 1
  Bi-racial/Multi-racial | 9 | 12 | 0 | 21

OUTCOME MEASURES:

1. Primary Outcome: The Pediatric Asthma Quality of Life Questionnaire (PAQOL)
Description: a 23-item instrument, 118 consists of three subdomains: activity limitation (5 items), emotional function (8 items), and symptoms (10 items). Higher scores indicate better levels of functioning. This scale has proved a valid and reliable measure of asthma-specific quality of life in adolescents. Mean scores are reported, and range from 1 to 7. Higher score indicating higher quality of life.
Time Frame: 15 months
Population: Number of participants analyzed included only those who had data collected at 15 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Number analyzed (Participants) | 139 | 124 | 27
score on a scale | 5.58 (1.36) | 5.93 (1.2) | 6.49 (0.85)
Statistical Analysis 1: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; For each model, partial eta squared (η2) was reported as the effect size for the change between treatment groups (Adult led vs. peer led asthma self-management). Partialη2 is the proportion of variance explained by a given variable out of the variance remaining after excluding variance explained by other predictors. Partial η2> 0.14 indicates large effects, while η2= 0.06 to 0.14 medium and < 0.06 small effects; Test type: Superiority; p = .043, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .003
Statistical Analysis 2: Comparison: Peer Leaders; For each model, partial eta squared (η2) was reported as the effect size for the overall change over time. Partialη2 is the proportion of variance explained by a given variable out of the variance remaining after excluding variance explained by other predictors. Partial η2> 0.14 indicates large effects, while η2= 0.06 to 0.14 medium and < 0.06 small effects; Test type: Superiority; p = .00, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .21
Statistical Analysis 3: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; Mediator analysis of AMI-SEI subscale on quality of life; Test type: Superiority; p = .0079, Sobel; Sobel Statistic = 2.4119
Statistical Analysis 4: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; Mediator analysis of ACQ Total score subscale on quality of life; Test type: Superiority; p = .0172, Sobel; Sobel Statistic = 2.1132

2. Secondary Outcome: Adolescent Asthma Knowledge Questionnaire (AAK)
Description: This 30-item instrument is a modification of the original 27-item questionnaire measuring children's knowledge of triggers and symptom identification and asthma management procedures. Total score range from 0 to 30, with higher score indicating greater knowledge.
Time Frame: 15 months
Population: Number of participants analyzed included only those who had data collected at 15 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Number analyzed (Participants) | 131 | 124 | 27
units on a scale | 23.07 (4.13) | 23.53 (4.16) | 25.85 (3.22)
Statistical Analysis 1: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.295, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .001
Statistical Analysis 2: Comparison: Peer Leaders; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .00, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .15

3. Secondary Outcome: Attitude Toward Asthma Scale (ATA)
Description: This 13-item scale measures children's attitudes toward their asthma on a 5-point Likert-type scale. Mean score ranges from 1 to 5, with higher score indicating a more positive attitude.
Time Frame: 15 months
Population: Number of participants analyzed included only those who had data collected at 15 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Number analyzed (Participants) | 136 | 124 | 27
score on a scale | 3.58 (0.73) | 3.77 (0.67) | 3.95 (0.74)
Statistical Analysis 1: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .140, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .002
Statistical Analysis 2: Comparison: Peer Leaders; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .00, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .15

4. Secondary Outcome: Asthma Self-Efficacy (ASE)
Description: This 14-item instrument measured on a 5-point scale (from 1='not at all sure' to 5='completely sure') assesses a child's confidence in attack prevention (e.g., learning asthma self-management skills, correct use of medication) and attack management (e.g., control symptoms, decide which medication to use). A total score was computed, ranging from 14 and 70, with higher values indicating greater self-efficacy.
Time Frame: 15 months
Population: Number of participants analyzed included only those who had data collected at 15 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Number analyzed (Participants) | 134 | 124 | 26
score on a scale | 56.38 (11.46) | 58.36 (11.79) | 63.62 (8.69)
Statistical Analysis 1: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .268, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .001
Statistical Analysis 2: Comparison: Peer Leaders; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .14, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .06

5. Secondary Outcome: Asthma Outcome Expectation Scale (AOE)
Description: This 5 items scale measured on a 9-point scale from 'not all all (1)' to 'extremely (9)' assess the construct of "outcome expectations" derived from social cognitive theory. The average score was computed, ranging from 1 to 9, with higher scores suggesting more positive expectations about performing actions of asthma self-management.
Time Frame: 15 months
Population: Number of participants analyzed included only those who had data collected at 15 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Number analyzed (Participants) | 135 | 124 | 27
units on a scale | 5.87 (1.38) | 6 (1.05) | 6.27 (1.13)
Statistical Analysis 1: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .238, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .001
Statistical Analysis 2: Comparison: Peer Leaders; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .43, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .03
Statistical Analysis 3: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; Test type: Superiority; p = .024, Mixed Models Analysis; Slope = -.203

6. Secondary Outcome: Asthma Prevention Index
Description: This is one of 3 subscales of asthma self-management indices developed for adolescents with asthma. The prevention index consists of 11 items measured on a 3-point scale. An average score based on items 1-9 was computed, ranging from 1 to 3, with higher scores suggesting greater regularity of prevention steps.
Time Frame: 15 months
Population: Number of participants analyzed included only those who had data collected at 15 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Number analyzed (Participants) | 136 | 124 | 27
score on a scale | 2.20 (0.51) | 2.11 (0.56) | 2.18 (0.62)
Statistical Analysis 1: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .484, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .000
Statistical Analysis 2: Comparison: Peer Leaders; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .00, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .12

7. Secondary Outcome: Asthma Management Index (AMI)
Description: This is one of the 3 subscales of Asthma Self-Management Indices. This subscale (9 items total) measures the number of steps taken to manage symptoms once they occur, and two response options are given, 0=no and 1=yes. Items 1-4, 6, 8 & 9 were summed for a total count of management steps taken, with possible scores ranging from 0 to 7. The higher the sum scores, the greater the number of steps taken to manage symptoms.
Time Frame: 15 months
Population: Number of participants analyzed included only those who had data collected at 15 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Number analyzed (Participants) | 136 | 124 | 27
score on a scale | 5.51 (1.54) | 5.67 (1.31) | 5.04 (1.97)
Statistical Analysis 1: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .648, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .000
Statistical Analysis 2: Comparison: Peer Leaders; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .04, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .07

8. Secondary Outcome: Asthma Management Self-efficacy Index
Description: This is one of 3 subscales of asthma self-management indices developed for adolescents with asthma. The self-efficacy index consists of 14 items measured on a 6-point scale (1='I am very sure I could not'; 6='I am very sure I could'). An average score of all 14 items was computed, ranging from 1 to 6, with higher scores suggesting greater self-efficacy.
Time Frame: 15 months
Population: Number of participants analyzed included only those who had data collected at 15 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Number analyzed (Participants) | 136 | 124 | 27
score on a scale | 4.79 (1.05) | 4.96 (0.85) | 5.40 (0.86)
Statistical Analysis 1: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .020, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .003
Statistical Analysis 2: Comparison: Peer Leaders; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .23, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .04

9. Secondary Outcome: Asthma Control Questionnaire (ACQ)
Description: ACQ consists of 6-items measuring asthma control based on the frequency, severity, and types of symptoms, as well as degree of activity limitation, and use of SABA in the past 7 days. Each item was responded on a 6-point scale from 0 to 6. Average scores were computed, with higher scores indicating worse asthma control.
Time Frame: 15 months
Population: Number of participants analyzed included only those who had data collected at 15 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
Number analyzed (Participants) | 139 | 124 | 27
score on a scale | 1.15 (1.01) | 0.92 (1.06) | 0.44 (0.64)
Statistical Analysis 1: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .049, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .002
Statistical Analysis 2: Comparison: Peer Leaders; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .00, Mixed Models Analysis — A priori threshold for statistical significance is <.05; partial eta squared = .12
Statistical Analysis 3: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; Test type: Superiority; p = .004, Mixed Models Analysis; Slope = -.294
Statistical Analysis 4: Comparison: Adult Led Asthma Self-Management vs Peer Led Asthma Self-Management; Mediator analysis of AMI-SEI subscale on ACQ total; Test type: Superiority; p = .0093, Sobel; Sobel Statistic = -2.3505

ADVERSE EVENTS:
Time Frame: Study time frame of 15 months from baseline to final follow up with participants.
Arm/Group | Adult Led Asthma Self-Management | Peer Led Asthma Self-Management | Peer Leaders
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/168 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/168 | 0/51
Other Adverse Events (participants affected / at risk) | 0/152 | 0/168 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT02293499/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2014-09-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT02293499/Prot_SAP_002.pdf